CLINICAL TRIAL: NCT07041021
Title: Effect of Intraoperative Fluid Management Guided by Respiratory Variations of Internal Jugular Vein on Postoperative Complications in Abdominal Surgeries: A Prospective Randomized Controlled Trial
Brief Title: Intraoperative Fluid Management Guided by Internal Jugular Vein on Postoperative Complications in Abdominal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohammad E Salama, MD, Principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5988#
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Complications
Keywords: Postoperative Complications; Abdominal surgeries; Internal Jugular Vein; Intraoperative fluid therapy
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Jugular Vein (IJV) group (Study group) (Active Comparator): In this group, fluid therapy will be guided by the respiratory variation of IJV throughout the surgery.
  Interventions: Diagnostic Test: Respiratory variation of the Internal Jugular Vein (IJV)
- Control group (No Intervention): In this group, conventional fluid therapy will be given to ensure that the mean arterial blood pressure is equal to or more than 65 mmHg.

INTERVENTIONS:
Diagnostic Test: Respiratory variation of the Internal Jugular Vein (IJV) — In the study group, the fluid therapy will be guided by the respiratory variation (RV) of the Internal Jugular Vein (IJV) throughout surgery. Fluid maintenance will be continued as long as the IJV diameter is less than 2 cm and the IJV RV is more than 18. If the IJV diameter exceeds 2 cm and the IJV RV is less than 18, fluids will be stopped.
  Arms: Internal Jugular Vein (IJV) group (Study group)

SUMMARY:
This study investigates the role of respiratory variation in the internal jugular vein as a tool for intraoperative fluid management during abdominal surgeries under general anesthesia.

The purpose of this clinical trial is to reduce postoperative complications and improve patient outcomes through proper intraoperative fluid management.

The main question it aims to answer is: Can intraoperative fluid management guided by the respiratory variation of the internal jugular vein during abdominal surgeries reduce postoperative complications? Research Hypothesis (Alternative Hypothesis): We hypothesize that fluid management guided by the respiratory variation of the internal jugular vein during abdominal surgeries can reduce postoperative complications.

The patients will be divided into two groups and randomized to receive either intraoperative fluid therapy guided by the respiratory variation of the internal jugular vein or standard fluid therapy. Postoperative complications, length of hospital stay, total amount of fluid administered intraoperatively, use of vasopressors in both groups, and incidence of hypotensive episodes will be recorded.

DETAILED DESCRIPTION:
Sonographic measurement of respiratory variation of IJV will be performed with a Philips CX50 ultrasound device (Philips Healthcare, Hamburg, Germany), equipped with a linear transducer. Respiratory variation of IJV will be measured by the same anesthesiologist with sufficient experience in ultrasound guided IJV cannulation. The anesthesiologist performing the ultrasound examinations will not be involved in this study and blinded to the hemodynamic parameters; a lead plate separated the monitor from the anesthesiologist and ultrasound device. The optimal short axis of the IJV will be obtained at the level of the cricoid cartilage by placement of the transducer perpendicular to the skin on the patient's neck in a transverse plane. The vein will be identified with color Doppler imaging as well as by compression. Ultrasound measurements will be performed on the left IJV, M-mode scan will be used to record the IJV diameter at the end of inspiration (IJVmax) and expiration (IJVmin) over an entire respiratory cycle. The images will be then frozen. The respiratory variation of IJV will be calculated with the following formula: IJV RV (%) = (IJVmax - IJVmin)/ (IJVmin) × 100%. The average values of IJVmax and IJVmin from three consecutive respiratory circles will be used in the analysis.

The finding of a small-diameter IJV (<1cm) and increased IJV RV (>18) suggest low-volume states. Conversely, a large IJV diameter (>2.1cm) and decreased IJV RV (<18) will suggest a high-volume state.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' American Society of Anesthesiologists physical status (ASA) is I and II.
2. The target age group is 20 to 70 years old.
3. Patients scheduled for abdominal surgery under general anesthesia with normal renal function.

Exclusion Criteria:

1. Refusal of the procedure or participation in the study.
2. Coagulopathy.
3. Pre-existing cardiac, renal, and respiratory diseases. 4-Internal jugular vein thrombosis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the incidence of postoperative complications in both groups, which will be measured by the occurrence of any of the postoperative complications during the first seven postoperative days in both groups | The first seven postoperative days
  Postoperative complications will include:
  (i) infections (urinary tract infection, wound infection, sepsis/septic shock) (ii) GI (Ileus, acute bowel obstruction, GI bleeding, abdominal compartment syndrome), (iii) Cardiovascular (deep venous thrombosis, pulmonary embolism, myocardial ischemia or infarction, cardiac arrest), (iv) Renal (AKI) (v) Respiratory (pneumonia, prolonged mechanical ventilation (more than 24 hours), respiratory failure, ARDS).

SECONDARY OUTCOMES:
The length of hospital stay in both groups | Up to 30 days postoperatively.
Assessment of the total amount of fluid administered intraoperatively in both groups | Intraoperatively (From the start to the end of the surgery)
Intraoperative vasopressor use in both groups | Intraoperatively (From the start to the end of the surgery)
Intraoperative hypotensive episodes in both groups | Intraoperatively (From the start to the end of the surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad E Salama, MD, Principal Investigator — Suez canal university hospitals
Locations (2):
- Egypt (2):
  - Suez Canal University Hospitals, Ismailia, Ismailia Governorate
  - Suez Canal University Hospitals, Ismailia

REFERENCES:
- [Background] Sanfilippo F, La Via L, Dezio V, Santonocito C, Amelio P, Genoese G, Astuto M, Noto A. Assessment of the inferior vena cava collapsibility from subcostal and trans-hepatic imaging using both M-mode or artificial intelligence: a prospective study on healthy volunteers. Intensive Care Med Exp. 2023 Apr 3;11(1):15. doi: 10.1186/s40635-023-00505-7. PMID 37009935
- [Background] Miller TE, Mythen M, Shaw AD, Hwang S, Shenoy AV, Bershad M, Hunley C. Association between perioperative fluid management and patient outcomes: a multicentre retrospective study. Br J Anaesth. 2021 Mar;126(3):720-729. doi: 10.1016/j.bja.2020.10.031. Epub 2020 Dec 13. PMID 33317803
- [Background] Ma GG, Hao GW, Yang XM, Zhu DM, Liu L, Liu H, Tu GW, Luo Z. Internal jugular vein variability predicts fluid responsiveness in cardiac surgical patients with mechanical ventilation. Ann Intensive Care. 2018 Jan 16;8(1):6. doi: 10.1186/s13613-017-0347-5. PMID 29340792
- [Background] Kan CFK, Skaggs JD. Current Commonly Used Dynamic Parameters and Monitoring Systems for Perioperative Goal-Directed Fluid Therapy: A Review. Yale J Biol Med. 2023 Mar 31;96(1):107-123. doi: 10.59249/JOAP6662. eCollection 2023 Mar. PMID 37009197
- [Background] Deslarzes P, Jurt J, Larson DW, Blanc C, Hubner M, Grass F. Perioperative Fluid Management in Colorectal Surgery: Institutional Approach to Standardized Practice. J Clin Med. 2024 Jan 30;13(3):801. doi: 10.3390/jcm13030801. PMID 38337495
- [Background] Dai S, Shen J, Tao X, Chen X, Xu L. Can ultrasonographic measurement of respiratory variability in the diameter of the internal jugular vein and the subclavian vein predict fluid responsiveness in parturients during cesarean delivery? A prospective cohort study. Heliyon. 2022 Dec 13;8(12):e12184. doi: 10.1016/j.heliyon.2022.e12184. eCollection 2022 Dec. PMID 36536919
- [Background] Kang D, Yoo KY. Fluid management in perioperative and critically ill patients. Acute Crit Care. 2019 Nov;34(4):235-245. doi: 10.4266/acc.2019.00717. Epub 2019 Nov 29. PMID 31795621
- [Background] Aaen AA, Voldby AW, Storm N, Kildsig J, Hansen EG, Zimmermann-Nielsen E, Jensen KM, Tibaek P, Mortensen A, Moller AM, Brandstrup B. Goal-directed fluid therapy in emergency abdominal surgery: a randomised multicentre trial. Br J Anaesth. 2021 Oct;127(4):521-531. doi: 10.1016/j.bja.2021.06.031. Epub 2021 Aug 11. PMID 34389168